CLINICAL TRIAL: NCT00765427
Title: A Phase 1a, Repeat-Dose Escalation Study to Investigate the Safety and Tolerability of a 7-Day Repeated Dose of Retinoid QLT091001 in Healthy Volunteers
Brief Title: Safety and Tolerability of Retinoid QLT091001 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: QLT Inc. (Industry)
Responsible Party: Sue-Anne Crocker, QLT Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: RET HV 01
Record Dates: First submitted 2008-09-30; First posted 2008-10-03 (Estimated); Last update posted 2009-03-30 (Estimated); Status verified 2009-03

CONDITIONS: Healthy Human Volunteers
MeSH Terms: interventions — retinol acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: QLT091001 — 7-day repeated dose

SUMMARY:
Healthy volunteer subjects will receive retinoid QLT091001 once-daily for 7 days for safety observation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects with ECG within normal limits and normal blood pressure and resting heart rate

Exclusion Criteria:

* Subjects with any clinically important abnormal physical finding at screening.
* Subjects who are actively participating in an experimental therapy study or who have received experimental therapy within 60 days of baseline.
* Female subjects who are either pregnant or lactating.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Clinical laboratory tests, ECG, vital signs, color vision, and visual acuity | 30 days

SECONDARY OUTCOMES:
Adverse events | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Victor Lao, MD, Principal Investigator; Andrew Strong, Ph.D., Study Director — QLT Inc.
Locations (1):
- Toronto, Ontario, Canada